CLINICAL TRIAL: NCT03560869
Title: Sympathetic Reactivity to Water Restriction in Young and Older Adults
Brief Title: The Effect of Acute Mild Dehydration on Blood Pressure Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 1097747; R01HL128388 (NIH); 5P20GM113125 (NIH)
Record Dates: First submitted 2018-06-06; First posted 2018-06-18 (Actual); Results first posted 2021-01-27 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Mild Dehydration
Keywords: Dehydration
MeSH Terms: conditions — Dehydration

STUDY DESIGN:
Intervention Model Description: Normal Hydration and Dehydration
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal hydration then dehydration (Experimental): Participants will consume water to maintain proper hydration for three days prior to testing (visit 1). Seven to 60 days later, participants will reduce water intake over three days and abstain from any water for the final 16 hours prior to testing (visit 2).
  Interventions: Other: Normal hydration; Other: Dehydration
- Dehydration than normal hydration (Experimental): Participants will reduce water intake over three days and abstain from any water for the final 16 hours prior to testing (visit 1). Seven to 60 days later, participants will consume water to maintain proper hydration for three days prior to testing (visit 2).
  Interventions: Other: Normal hydration; Other: Dehydration

INTERVENTIONS:
Other: Normal hydration — see description in 'arms'
Other: Dehydration — see description in 'arms'

SUMMARY:
The goal of this project is determine how acute mild dehydration impacts blood pressure control at rest and during static exercise. This protocol will test healthy young and older adults in a normally hydrated and dehydrated condition.

DETAILED DESCRIPTION:
The purpose of this project is determine how acute mild dehydration impacts blood pressure control at rest and during static exercise. Additionally, we will determine whether or not the sympathetic nervous system has a role in mediating blood pressure control at rest and during static exercise. This protocol will test healthy young and older adults in a normally hydrated and dehydrated condition. This will allow for a within participant comparison. Additionally, we will later determine if age alters blood pressure control at rest or during static exercise.

ELIGIBILITY:
Inclusion Criteria (Young):

• age: 20-35 years old

Exclusion Criteria (Young):

* high blood pressure (>140/90 mmHg)
* history of cardiovascular disease
* history of cancer
* history of diabetes
* history of kidney disease
* obesity (BMI > 30 kg/m2)
* smoking or tobacco use
* current pregnancy
* nursing mothers
* communication barriers

Inclusion Criteria (Older):

* age: 60-75 years old
* ECG within normal limits
* screening blood panel within normal limits

Exclusion Criteria (Older):

* high blood pressure (>140/90 mmHg)
* history of cardiovascular disease
* history of cancer
* history of diabetes
* history of kidney disease
* obesity (BMI > 30 kg/m2)
* smoking or tobacco use
* current pregnancy
* nursing mothers
* communication barriers

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-08-08 (Actual); Primary Completion 2019-06-13 (Actual); Study Completion 2019-06-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- William B Farquhar, Newark, Delaware, United States

REFERENCES:
- [Result] Watso JC, Robinson AT, Babcock MC, Migdal KU, Wenner MM, Stocker SD, Farquhar WB. Short-term water deprivation does not increase blood pressure variability or impair neurovascular function in healthy young adults. Am J Physiol Regul Integr Comp Physiol. 2020 Jan 1;318(1):R112-R121. doi: 10.1152/ajpregu.00149.2019. Epub 2019 Oct 16. PMID 31617739
- [Result] Watso JC, Babcock MC, Robinson AT, Migdal KU, Wenner MM, Stocker SD, Farquhar WB. Water deprivation does not augment sympathetic or pressor responses to sciatic afferent nerve stimulation in rats or to static exercise in humans. J Appl Physiol (1985). 2019 Jul 1;127(1):235-245. doi: 10.1152/japplphysiol.00005.2019. Epub 2019 May 9. PMID 31070954
- [Result] Robinson AT, Babcock MC, Watso JC, Brian MS, Migdal KU, Wenner MM, Farquhar WB. Relation between resting sympathetic outflow and vasoconstrictor responses to sympathetic nerve bursts: sex differences in healthy young adults. Am J Physiol Regul Integr Comp Physiol. 2019 May 1;316(5):R463-R471. doi: 10.1152/ajpregu.00305.2018. Epub 2019 Feb 22. PMID 30794437

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants completed both conditions.
Groups:
- Normal Hydration Than Dehydration: 14 participants consumed water to maintain proper hydration for three days prior to testing (visit 1). Seven to 60 days later, participants reduced water intake over three days and abstained from any water for the final 16 hours prior to testing (visit 2).
- Dehydration Than Normal Hydration: 21 participants reduced water intake over three days and abstained from any water for the final 16 hours prior to testing (visit 1). Seven to 60 days later, participants consumed water to maintain proper hydration for three days prior to testing (visit 2).
Period: Overall Study
Arm/Group | Normal Hydration Than Dehydration | Dehydration Than Normal Hydration
Started | 14 | 21
Completed | 7 | 12
Not Completed | 7 | 9
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Screening failure | 4 | 4
Not completed — Withdrawal by PI | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All Study Participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 28
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Blood Pressure Variability
Description: Blood pressure variability (BPV) was calculated using standard deviation and using the average real variability index of blood pressure values. The average real variability index calculates the average of absolute differences between consecutive BP measurements and is thought to provide further prognostic value compared with traditional measures of BPV.
Time Frame: During experimental visits 1 and 2
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Normal Hydration: Participants will consume water to maintain proper hydration for three days prior to testing.
  Hydration State: Hydration State
- Dehydration: Participants will reduce water intake over three days and abstain from any water for the final 16 hours prior to testing.
  Hydration State: Hydration State
Arm/Group | Normal Hydration | Dehydration
Number analyzed (Participants) | 19 | 19
mmHg | 2.6 (1.1) | 2.5 (0.9)

2. Primary Outcome: Blood Pressure Reactivity - Handgrip Exercise
Description: Change in systolic blood pressure during the second-minute handgrip exercise minus compared to pre-exercise baseline (i.e., at rest).
Time Frame: During experimental visits 1 and 2
Population: 4 adults were excluded from this analysis due to technical difficulties
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Normal Hydration | Dehydration
Number analyzed (Participants) | 15 | 15
mmHg | 20 (11) | 18 (8)

ADVERSE EVENTS:
Time Frame: Adverse event data were monitored throughout the study (during experimental protocol #1 (3 days), study visit #1 (1 day), washout (up to 60 days), experimental protocol #2 (3 days), study visit #2 (1 day), and the week (7 days) following this final study visit - i.e., up to 75 days).
Description: There were no adverse events, thus, there are no adverse event outcomes reported.
Arm/Group | Normal Hydration | Dehydration
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 0/35 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2018-07-19): https://cdn.clinicaltrials.gov/large-docs/69/NCT03560869/ICF_000.pdf
  • Study Protocol (2019-03-06): https://cdn.clinicaltrials.gov/large-docs/69/NCT03560869/Prot_001.pdf